CLINICAL TRIAL: NCT05563896
Title: The Energy Cost of Living in the Developing World
Status: Completed | Type: Observational
Sponsor: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Collaborators: University Cheikh Anta Diop of Daka (Unknown); Tehran University of Medical Sciences (Other); University of Aberdeen (Other); Tohoku University (Other); Moi University (Other)
Responsible Party: Principal Investigator, John R. Speakman, Principal Investigator, Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Other Study IDs: SIAT-IRB-220715-H0604
Record Dates: First submitted 2022-09-25; First posted 2022-10-03 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Food Requirements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- China: We plan to enroll 200 healthy adults in this study at five different international sites (China, Iran, Kenya, Senegal, UAE). Forty subjects will be enrolled at each site. Previous studies showed energy requirements varied with sex and age of the participants. Therefore, in each site, 20 males and 20 females will be recruited respectively. The samples will comprise individuals aged 18-50. Half will be male and half female. Half of the samples will be collected in 'summer' (June, July and August) and half in 'winter' (October, November and December). The same individuals will not be measured in both seasons.
  Interventions: Other: No intervention
- Sénégal: Forty subjects will be enrolled at Senegal site.In Senegal site, 20 males and 20 females will be recruited respectively. The samples will comprise individuals aged 18-50. Half will be male and half female. Half of the samples will be collected in 'summer' (June, July and August) and half in 'winter' (October, November and December). The same individuals will not be measured in both seasons.
  Interventions: Other: No intervention
- Kenya: Forty subjects will be enrolled at Kenya site.In Kenya site, 20 males and 20 females will be recruited respectively. The samples will comprise individuals aged 18-50. Half will be male and half female. Half of the samples will be collected in 'summer' (June, July and August) and half in 'winter' (October, November and December). The same individuals will not be measured in both seasons.
  Interventions: Other: No intervention
- Iran: Forty subjects will be enrolled at Iran site.In Iran site, 20 males and 20 females will be recruited respectively. The samples will comprise individuals aged 18-50. Half will be male and half female. Half of the samples will be collected in 'summer' (June, July and August) and half in 'winter' (October, November and December). The same individuals will not be measured in both seasons.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
By 2050 there will be 9 billion people on earth. Yet a major issue facing governments is that the current method by which food demands are estimated is widely acknowledged to be completely inaccurate. There is an accurate method available. It is based on measurements of isotope elimination and is called the doubly-labeled water (DLW) method. As part of an initiative sponsored by the International Atomic energy agency (IAEA), the investigators recently compiled a database of measurements using this technique. It showed that use of the DLW method has been mostly restricted to the USA and western Europe. It has been rarely applied across Africa and Asia. There is a clear need to fill this gap in our knowledge providing information that governments across the belt and road countries can use to forecast future food demands. A letter of support from the IAEA confirms the practical importance of having these data which will become reference standards for food intake estimates across the region. Having this information not only fills a very practical need, but also has a strong scientific purpose. The population of earth is not only getting bigger, but the people are getting fatter. The causes of this obesity epidemic are strongly disputed with some suggesting it is due to our increasingly sedentary lives (computers, cars, phones etc), but others suggesting it is mostly due to changing food patterns (junk food and sugar sweetened beverages). Measuring energy expenditure of people across countries that vary enormously in their levels of obesity will address whether falling expenditure due to lowered physical activity is a key cause of the epidemic.

DETAILED DESCRIPTION:
Energy Expenditure and Activity

Energy expenditure, body composition, and metabolism will be assessed by the following measures:

Total Energy Expenditure (TEE) using Doubly-labeled water (DLW):

TEE will be measured using the DLW method. Urine samples from all participants in the DLW subset will be stored at -20 oC and shipped on dry ice for analysis in the laboratory of Dr. John Speakman at the University of Aberdeen, or the Shenzhen Institute of Advanced Technology, Chinese academy of sciences. Isotopes will be measured in benchtop near-infrared isotope gas analyzer, and mean CO2 production will be calculated from isotope ratios using the recently derived equation. TEE will then be calculated using mean CO2 production.

Resting Metabolic Rate (RMR):

RMR will be measured by indirect calorimetry while participants are resting supine in thermoneutral conditions. Oxygen consumption and CO2 production will be measured over a period of 25 min, and measurements from the final 10 min will be used to calculate RMR using Weir's equation. Calorimeters will be assessed with a turbine test to ensure accuracy of measurements.

Physical Activity:

Physical activity estimates obtained from the activity monitors will be used to assess energy expenditure concurrently with TEE and RMR measurements. The output generated from the accelerometer worn near the hip will include the following: 24-hour physical activity and sleep/wake measurements including acceleration, activity counts, energy expenditure, and physical activity intensity.

Body Composition

Bioelectrical impedance (BIA):

The BIA method will be used to estimate total body water, fat and fat free mass using the BIA machine available at each site. Since this is a cross-sectional study, a uniform BIA machine is not specified as a requirement in the protocol. Where available body composition by DZ=XA will also be measured.

Height, Weight, Waist Circumference, and Blood Pressure:

Duplicate measurements of weight (to +0.1kg), height (to +0.1 cm), hip and waist circumference (to +0.3 cm), and blood pressure will be taken. At visit 1, fasting weight will be measured at the beginning of the visit. Fasting weight will be measured at visit 2 and, if applicable.

Environmental temperature:

The Ibutton (DS1921G) monitors will be provided for the assessment of both indoor and outdoor temperature of their living environment. The iButtons can be affixed to the handbag (or clothes) to measure the subject exposure temperature, an indoor wall of home and workplace, and the building outside to measure the outdoor temperature using a strip of adhesive, water resistant, medical grade tape.

Metabolomics and SNP genotyping:

The subjects will have their venous blood collected in a fasted state. 4ml of venous blood (BD vacutainer K2 EDTA, BD, USA) will be used to separate plasma for metabolomics analysis and to extract genomic DNA (TIANamp Blood DNA kit, TIANGEN, China. QIAamp Midi Blood DNA kit, QIAGEN, Germany) for Single nucleotide polymorphism (SNP) genotyping (Agena MassARRAY, CapitalBio Technology, China).

ELIGIBILITY:
Inclusion Criteria:

* adults working at least 3 out of 7 days per week for a total of >12 hours per week
* ages 18-50 years
* willing to enroll in the study and complete all study requirements

Exclusion Criteria:

* current pregnancy or pregnancy within the last 12 months, and/or currently breast feeding or lactating
* Individuals with known non-communicable disease notably diabetes, cardiovascular disease or cancer
* any diseases or chronic use of medications that would influence ability to comply with the study requirements
* Individuals with infectious disease will also be excluded (HIV, Lassa fever, malaria and Sars-Cov2) In sites where large populations adhere to Ramadan, we will avoid religious festival periods.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 200 healthy adults will be enrolled in this study at five different international sites (China, Iran, Kenya, Senegal, UAE). Forty subjects will be enrolled at each site. In each site, 20 males and 20 females will be recruited respectively. The samples will comprise individuals aged 18-50. Half will be male and half female. Half of the samples will be collected in 'summer' and half in 'winter'. The same individuals will not be measured in both seasons. Once enrollment goals for the subsets have been reached, incoming participants will no longer be offered the opportunity to participate in the project.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Total Energy Expenditure (TEE) | 14 days
  TEE will be measured using the DLW method. Urine samples from all participants in the DLW subset will be stored at -20 oC and shipped on dry ice for analysis in the laboratory of Dr. John Speakman at the University of Aberdeen, or the Shenzhen Institute of Advanced Technology, Chinese academy of sciences. Isotopes will be measured in benchtop near-infrared isotope gas analyzer, and mean CO2 production will be calculated from isotope ratios using the recently derived equation. TEE will then be calculated using mean CO2 production.
Resting Metabolic Rate (RMR) | 40 minutes
  RMR will be measured by indirect calorimetry while participants are resting supine in thermoneutral conditions. Oxygen consumption and CO2 production will be measured over a period of 25 min, and measurements from the final 10 min will be used to calculate RMR using Weir's equation. Calorimeters will be assessed with a turbine test to ensure accuracy of measurements.
Physical Activity | 14 days
  Physical activity estimates obtained from the activity monitors will be used to assess energy expenditure concurrently with TEE and RMR measurements. The output generated from the accelerometer worn near the hip will include the following: 24-hour physical activity and sleep/wake measurements including acceleration, activity counts, energy expenditure, and physical activity intensity
Bioelectrical impedance | 10 minutes
  The BIA method will be used to estimate total body water, fat and fat free mass using the BIA machine available at each site. Since this is a cross-sectional study, a uniform BIA machine is not specified as a requirement in the protocol. Where available body composition by DZ=XA will also be measured.
Height, Weight, Waist Circumference, and Blood Pressure | 20 minutes
  Duplicate measurements of weight (to +0.1kg), height (to +0.1 cm), hip and waist circumference (to +0.3 cm), and blood pressure will be taken. At visit 1, fasting weight will be measured at the beginning of the visit. Fasting weight will be measured at visit 2 and, if applicable.
Environmental temperature | 14 days
  The Ibutton (DS1921G) monitors will be provided for the assessment of both indoor and outdoor temperature of their living environment. The iButtons can be affixed to the hand bag (or clothes) to measure the subject exposure temperature, an indoor wall of home and workplace, and the building outside to measure the outdoor temperature using a strip of adhesive, water resistant, medical grade tape.

SECONDARY OUTCOMES:
Metabolomics | 1 month
  The subjects will have their venous blood collected in a fasted state. 4ml of venous blood (BD vacutainer K2 EDTA, BD, USA) will be used to separate serum for metabolomics analysis. The subjects will have their faecal samples collected by penkit and extract the microbial DNA for Microbiomics analysis. Serum microbiome DNA samples will be shipped to Japan to get metabolomics analysed.
Microbiomics | 1 month
  The subjects will have their faecal samples collected by penkit and extract the microbial DNA for Microbiomics analysis. Faecal microbiome DNA samples will be shipped to Japan to get Microbiomics analysed.

CONTACTS AND LOCATIONS:
Overall Officials: John R. Speakman, Doctor, Principal Investigator — Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Locations (1):
- Shenzhen Institute of Advanced Technology,Chinese Academy of Sciences, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Speakman JR, Yamada Y, Sagayama H, Berman ESF, Ainslie PN, Andersen LF, Anderson LJ, Arab L, Baddou I, Bedu-Addo K, Blaak EE, Blanc S, Bonomi AG, Bouten CVC, Bovet P, Buchowski MS, Butte NF, Camps SGJA, Close GL, Cooper JA, Creasy SA, Das SK, Cooper R, Dugas LR, Ebbeling CB, Ekelund U, Entringer S, Forrester T, Fudge BW, Goris AH, Gurven M, Hambly C, El Hamdouchi A, Hoos MB, Hu S, Joonas N, Joosen AM, Katzmarzyk P, Kempen KP, Kimura M, Kraus WE, Kushner RF, Lambert EV, Leonard WR, Lessan N, Ludwig DS, Martin CK, Medin AC, Meijer EP, Morehen JC, Morton JP, Neuhouser ML, Nicklas TA, Ojiambo RM, Pietilainen KH, Pitsiladis YP, Plange-Rhule J, Plasqui G, Prentice RL, Rabinovich RA, Racette SB, Raichlen DA, Ravussin E, Reynolds RM, Roberts SB, Schuit AJ, Sjodin AM, Stice E, Urlacher SS, Valenti G, Van Etten LM, Van Mil EA, Wells JCK, Wilson G, Wood BM, Yanovski J, Yoshida T, Zhang X, Murphy-Alford AJ, Loechl CU, Melanson EL, Luke AH, Pontzer H, Rood J, Schoeller DA, Westerterp KR, Wong WW; IAEA DLW database group. A standard calculation methodology for human doubly labeled water studies. Cell Rep Med. 2021 Feb 16;2(2):100203. doi: 10.1016/j.xcrm.2021.100203. eCollection 2021 Feb 16. PMID 33665639
- [Background] WEIR JB. New methods for calculating metabolic rate with special reference to protein metabolism. J Physiol. 1949 Aug;109(1-2):1-9. doi: 10.1113/jphysiol.1949.sp004363. No abstract available. PMID 15394301